CLINICAL TRIAL: NCT06738446
Title: Multicomponent Dietary Supplementation: Impact on Tear Secretion and Ocular Surface Inflammation in Dry Eye Syndrome Patients
Brief Title: Dietary Supplementation on Tear Secretion and Inflammation in DES
Acronym: DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shih Chien Huang (Other)
Collaborators: Far East Bio-Tec Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Shih Chien Huang, Assistant Professor, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSI-20199
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye Syndrome (DES)
Keywords: Dry eye syndrome; inflammation; oxidative stress; fish oil; lutein; zeaxanthin
MeSH Terms: conditions — Dry Eye Syndromes; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): This group is used only as a control.
- Multicomponent Dietary Supplement group (Experimental): 45 mg/day EPA, 30 mg/day DHA, 30 mg/day lutein, and 1.8 mg/day zeaxanthin
  Interventions: Dietary Supplement: Multicomponent dietary supplement group

INTERVENTIONS:
Dietary Supplement: Multicomponent dietary supplement group — Participants in supplement group were asked to take a capsule content are eicosapentaenoic acid 45 mg, docosahexaenoic acid 30 mg, lutein 30 mg, and zeaxanthin1.8 mg every day for 12 weeks
  Arms: Multicomponent Dietary Supplement group

SUMMARY:
The goal of this clinical trial is to explore the effect of supplementation of fish oil, lutein and zeaxanthin on the symptoms of dry eye syndrome, antioxidant capacity, oxidative stress and anti-inflammatory capacity in DES patients., it aims to answer are:

To evaluate the effects of a 12-week multicomponent dietary supplementation (capsule content are eicosapentaenoic acid 45 mg, docosahexaenoic acid 30 mg, lutein 30 mg, and zeaxanthin1.8 mg)on symptoms of dry eye syndrome, oxidative stress, antioxidant capacity, and inflammation.

To investigate the relationships between dry eye symptoms, oxidative stress, antioxidant capacity, and inflammation.

Participants will be randomly assigned to control group (n = 50) and supplement group (n = 50) and white pomegranate extract group (n = 50) for 12 weeks. Participants will complete assessments of tear secretion, antioxidant capacity, and ocular surface inflammation.

DETAILED DESCRIPTION:
1. Study Participants i. Inclusion criteria: (1) Aged 20 to 80 years; (2) Diagnosed with moderate or greater dry eye syndrome by an ophthalmologist.

   ii. Exclusion criteria: Previous ocular surgery within the last 3 months. iii. Withdrawal Criteria Participants are free to decide whether to participate in this trial, and they can withdraw their consent at any time during the trial without providing any reason. If participants experience discomfort, they may withdraw from the trial at any time without facing any penalties or compromising their rights.

   iv. Participants were randomly assigned to a supplement group or control group. Participants in supplement group were asked to take a capsule content are eicosapentaenoic acid 45 mg, docosahexaenoic acid 30 mg, lutein 30 mg, and zeaxanthin1.8 mg every day for 12 weeks.
2. Subject Recruitment Interested participants will be recruited openly through posters posted at Chung Shan Medical University Hospital. The researchers will explain the trial content for 15-20 minutes, and if interested, participants will sign the informed consent form.
3. Research Methods At weeks 0 and 12 of the trial, 10 μL of tear samples and 10 mL of blood samples will be collected from participants.

   i. The basic and OSDI questionnaires and ii. Evaluate dry eye-related indicators evaluation iii. Measure blood or tear oxidative stress and antioxidant capacity, and tear inflammatory factors were measured.
4. All statistical data will be analyzed using SigmaPlot statistical software (version 12.5; Systat Software, San Jose, CA), and the data will be presented using an intention-to-treat (ITT) approach. The differences in continuous data between the two groups will be compared using the Student's t-test. The differences in values within the group before and after intervention will be compared using the paired t-test. The differences in ordinal data between the two groups will be assessed using the Chi-square test. Partial Spearman's correlation will be used to adjust for confounding factors (age, gender, and menopause status) to explore the correlations between changes in oxidative stress and antioxidant capacity in blood and tears, changes in inflammatory factors, and changes in dry eye assessment. Multiple linear regression will be used to analyze the effect of supplement intake on changes in oxidative stress and antioxidant capacity in blood and tears, changes in inflammatory factors, and changes in dry eye assessment. The data will be expressed as mean ± standard deviation (SD), with p < 0.05 indicating statistical significance.

Through this study, the administration of multicomponent dietary supplementation to patients with dry eye syndrome aims to understand whether different eye health nutrients improve tear secretion, antioxidant capacity, and anti-inflammatory responses. This may serve as an adjunctive treatment or symptom relief for dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 20 and 80 years,
2. moderate or above severity of dry eye syndrome.

Exclusion Criteria:

1. undergoing ophthalmic surgery within the past three months,
2. autoimmune diseases,
3. ocular allergies,
4. consumption of fish oil or antioxidant supplements within the past three months, and
5. pregnant or lactating women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | 12 weeks
  We aim to improve the symptoms of dry eye disease in patients by administering dietary supplements

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chien Huang, Dr, Study Chair — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan